CLINICAL TRIAL: NCT01128660
Title: Assessment of the Prescriber's and the Pharmacies Overview of Patient Medication by Use of the Fidelity Coefficient.
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jesper Hallas, Professor of Clinical Pharmacology, University of Southern Denmark
Other Study IDs: JH-AP-001
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Misuse of Prescription Only Drugs
Keywords: Prescription, General practitioner, Pharmacy
MeSH Terms: conditions — Prescription Drug Misuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RSD-citizens: Residents of Southern Denmark, who filed more than 9 prescriptions during 2009.

SUMMARY:
The purpose of this study is to twofold. The investigators wish to introduce a new patient-descriptive parameter, the 'Fidelity Coefficient', and use it to assess and compare the overview of patient's medication possessed by the general practitioners and the pharmacies.

DETAILED DESCRIPTION:
The fidelity coefficient, FC, is a measure of what proportion of individual patients' medication that are accounted for by the most used prescriber and the most used pharmacy. Each patient therefore has two values, one describing his fidelity towards his most used prescriber, FCPresc, and one describing his fidelity towards his most used pharmacy, FCPharm.

The investigators intend to assess this parameter in an observational population scale database study, using standard descriptive statistics, and subsequently compare the obtained average FCPresc and FCPharm.

Furthermore, the investigators will analyze the two obtained FCs for dependency of a predefined list of variables: age, gender, number of prescriptions, whether the most frequent prescriber was a GP and whether the most used pharmacy was urban.

Finally, the investigators intend to analyze which medications (grouped using the ATC-system with 4 digits, e.g. C07A) that has the highest proportion of prescriptions that were either issued by a non-main prescriber or redeemed at a non-main pharmacy, which roughly translates into the most 'infidel' medications. To insure relevance we intend to use a cut-off-value of the medication being prescribed at least 50.000 times, which equals about 85 % of the data according to preceding analyses.

The data for this study will be obtained from the Odense University Pharmacoepidemiological Database (OPED). In brief, it is a research database with full coverage of all reimbursed prescriptions in the Region of Southern Denmark (1.2 million inhabitants). The data included in each prescription record includes the prescription holder, the prescriber, the pharmacy, the date of dispensing and a full account of the dispensed product, including substance, brand name, route of administration, ATC-code and Defined Daily Dose (DDD).

Some drugs are exempt from re-imbursement and thus not covered by the database, including benzodiazepines, oral contraceptives, laxatives and certain antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Having filed more than 9 prescriptions during 2009.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Region of Southern Denmark during 2009.
Sampling Method: Probability Sample
Enrollment: 283388 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
FC(Pharm) | cross-sectional study with data aquisition over one year
  The pharmacy fidelity coefficient, FC(Pharm), is a measure of what proportion of individual patients' medication that are accounted for by the most used pharmacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Hallas, MD, PhD, Principal Investigator — Professor, Research Unit of Clinical Pharmacology, University of Southern Denmark.; Anton Pottegard, BSc in Pharm, Principal Investigator — Guest Researcher, Research Unit of Clinical Pharmacology, University of Southern Denmark.
Locations (1):
- Research Unit of Clinical Pharmacology, University of Southern Denmark, Odense, Funen, Denmark

REFERENCES:
- [Background] Pottegard A, Hallas J. Physicians' and pharmacies' overview of patients' medication. An analysis of fidelity coefficients. Eur J Clin Pharmacol. 2011 Sep;67(9):919-24. doi: 10.1007/s00228-011-1026-3. Epub 2011 Mar 12. PMID 21399945